CLINICAL TRIAL: NCT01640600
Title: Yale Pink and Blue Kids: Effects of in Utero Exposure to Nicotine and Selective Serotonin Reuptake Inhibitors in 4-8 Year Old Children
Brief Title: Yale Pink and Blue Kids: Effects of Exposure During Pregnancy to Nicotine or Antidepressants in 4-8 Year Old Children
Acronym: PABKids
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1105008516
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2016-12

CONDITIONS: Behavioral Problems; Cognitive Problems; Motor Development
Keywords: To determine whether 4-8 year-old children exposed to nicotine or antidepressants in utero have more behavioral problems.; To determine whether 4-8 year-old children exposed to nicotine or antidepressants in utero have more cognitive problems.; To determine whether 4-8 year-old children exposed to nicotine or antidepressants in utero have poorer motor development.
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — We will be collecting saliva from mothers and their children in order to look at certain genes that may be related to developmental outcomes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Children exposed to SSRIs in utero: This group are comprised of children whose mothers used antidepressants during pregnancy and who were therefore exposed to antidepressants in utero.
- Children exposed to nicotine in utero: This group is comprised of children whose mothers smoked cigarettes during pregnancy and who were therefore exposed to nicotine in utero.
- Children exposed to neither nicotine nor SSRIs: This group is comprised of children who were exposed to neither nicotine nor SSRIs in utero.

SUMMARY:
The purpose of this project is to conduct a follow-up study with women that had participated in the Yale Pink and Blue Study of depression in pregnancy and birth outcomes. The Yale Pink and Blue Kids Study is a follow-up study with the mothers and also with the children they were pregnant with in Yale Pink and Blue. These children are now between the ages of 4 and 8 years old, which is a perfect time to look at developmental outcomes in children. This study will look at children with exposure to nicotine or antidepressants during pregnancy, as well as children who were not exposed. The investigators hypothesis is that children who were exposed to either nicotine or antidepressants in pregnancy will have poorer developmental outcomes than children who were not exposed. The investigators are also interested in determining whether nicotine exposure or antidepressant exposure results in poorer outcomes.

The investigators specific aims are:

1. To determine whether pre-school and school aged offspring exposed to maternal cigarette smoking or antidepressants during pregnancy are more likely to have social-emotional problems compared to children who were not exposed to cigarettes or antidepressants during pregnancy.
2. To determine whether pre-school and school aged children who were exposed to prenatal maternal cigarette smoking or antidepressants during pregnancy display cognitive impairments as compared to children who were not exposed to either prenatal maternal cigarette smoking or antidepressants.
3. To determine if pre-school and school aged children who were exposed to maternal prenatal cigarette smoking or antidepressants display impaired motor development as compared to children who were not exposed to maternal cigarette smoking or antidepressants in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the Yale Pink and Blue Study and had children born between 2005 and 2008.
* Exposure to SSRIs during pregnancy will be defined as those women with no exposure in pregnancy and continuous use of SSRIs (defined as taking at least one SSRI during every trimester).
* Exposure to nicotine will be defined as no exposure (no cigarettes during pregnancy), light exposure (an average of less than one cigarette a day over pregnancy duration), and heavy exposure (an average of one cigarette a day over the duration of pregnancy.

Exclusion Criteria:

* Spanish-Speaking women and women who live over a one hour driving distance from Yale will be considered ineligible.
* Children are not eligible if their mother had gestational exposure to prescription drugs in the FDA-defined category of D or X, since this can confound our assessment.
* Women with discontinuous use of SSRIs (defined as using SSRIs during pregnancy, but not every trimester) will also be excluded.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each subject is a previous study participant known to this research team who has agreed to be contacted about future studies. We will review only their research records and not medical records in order to determine eligibility. There are no subjects for whom the ability to give informed consent can be questioned. All of the subjects were at least the age of 18 at the time of their initial PAB participation between 2005-2008, and thus are at least age 20 at the present time. All subjects are English speaking.
  These are women who participated in the PAB Study (HIC #12394) and delivered a singleton birth (no twins or triplets) between 2005-2008. We are inviting them and their children (now aged 4-8) to participate.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Externalizing and internalizing behavior | 1 year
  The Revised Child Behavior Checklist (CBCL-2) is one of the most widely-used measures for evaluating maladaptive behavioral and emotional problems in children between the ages of 2 and 18. It assesses internalizing (i.e., anxious, depressive, and overcontrolled) and externalizing (i.e., aggressive, hyperactive, noncompliant, and undercontrolled) behaviors. In addition to the CBCL-2, we will use direct observation of a 2-minute mother-child interaction session to measure externalizing and internalizing symptoms, as parent report on the CBCL-2 may be biased by maternal psychopathology.
Cognitive Impairment | 1 year
  Cognitive impairment is measured using the Kaufman Brief Intelligence Test (KBIT-2), which measures both verbal and nonverbal intelligence through questions , riddles, and pictures. A computer test, CogState, will also assess cognitive functioning, specifically executive functioning through card-related tasks that will ask a child to respond in different ways.
Fine & Gross Motor Development | 1 Year
  Fine and Gross Motor Skills will be measured using the Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) (10), the most widely administered test of fine and gross motor skills in children ages 4 to 21. Administration time is approximately 60 minutes. Subtests include: Fine Motor Precision, Fine Motor Integration, Manual Dexterity, and Bilateral Coordination.

CONTACTS AND LOCATIONS:
Overall Officials: Megan V Smith, DrPH, Principal Investigator — Yale University
Locations (1):
- Yale Psychiatry: The PMS, Perinatal, and Postpartum Research Program, New Haven, Connecticut, United States